CLINICAL TRIAL: NCT04517422
Title: Efficacy and Safety of Lactobacillus Plantarum and Pediococcus Acidilactici as Co-adjuvant Therapy for Reducing the Risk of Severe Disease in Adults With SARS-CoV-2 and Its Modulation of the Fecal Microbiota: A Randomized Clinical Trial
Brief Title: Efficacy of L. Plantarum and P. Acidilactici in Adults With SARS-CoV-2 and COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Collaborators: Innovacion y Desarrollo de Estrategias en Salud (Other); Hospital General Dr. Manuel Gea González (Other Government); Hospital Angeles del Pedregal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ABB-COVID19
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV Infection
Keywords: probiotics; sars-cov-2; covid-19; adults
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trials. 300 subjects (18-60 years old) will be allocated to receive a combination of Lactobacillus plantarum CECT 30292, Lactobacillus plantarum CECT 7484, Lactobacillus plantarum CECT 7485, and P. acidilactici CECT 7483 (branch one) or placebo (branch two)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study staff, including the Principal Investigator and the persons performing the subject assessments, will be blinded during the study. Sealed individual treatment code envelopes will be kept at the clinic to be able to break the code if any emergency occurs, as judged by the Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Active test product contains four lactic acid bacteria strains with Qualified Presumption of Safety (QPS)status by European Food Safety Authority (EFSA): Lactobacillus plantarum CECT30292, Lactobacillus plantarum CECT7484, Lactobacillus plantarum CECT7485, and Pediococcus acidilactici CECT7483, with maltodextrin (E1400, qs) as excipient, formulated in a vegetable hydroxymethylpropyl-cellulose capsule (HPMC) of size 0. Active test product is a food supplement and not an investigational medicinal product
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): The control study product is identical in packaging and formulation except that Lactobacillus plantarum CECT30292, Lactobacillus plantarum CECT7484, Lactobacillus plantarum CECT7485, and Pediococcus acidilactici CECT7483 (probiotic bacteria) are not present. The Control product only contains maltodextrin (E1400, qs) in a vegetable hydroxymethylpropyl-cellulose capsule (HPMC) of size 0.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Combination of Lactobacillus plantarum CECT30292, Lactobacillus plantarum CECT 7484, Lactobacillus plantarum CECT 7485, and Pediococcus acidilactici CECT 7483
  Arms: Probiotics
Other: Placebo — Combination of maltodextrin (E1400, qs) in a vegetable hydroxymethylpropyl-cellulose capsule (HPMC) of size 0
  Arms: Placebo

SUMMARY:
Clinical research focused to evaluate the effect as coadyuvant of a combination of L. plantarum and P. acidilactici in adults positive for SARS-CoV-2 with mild clinical COVID-19 symptoms. Main objective is to evaluate how this combination of probiotics reduce the risk to progress to moderate or severe COVID and associated advantages such as reduce the risk of death. Adittionnally this RCT is launching to explore the benefits of this combination of strains to modulate fecal microbiome and explore how this correlate with clinical improvement.

DETAILED DESCRIPTION:
Randomized controlled trial (RCT) to evaluate safety and efficacy of Lactobacillus plantarum CECT 30292, Lactobacillus plantarum CECT 7484, Lactobacillus plantarum CECT 7485 y P. acidilactici CECT 7483, one dose a day to reduce the risk of subjects with mild COVID-19 to evolute to moderate or severe disease. As secondary aims this trial is intented to evaluate the effect of this strains combinations to reduce the frequency and severity of gastrointestinal COVID-19 symptoms and lung abnormalities, to reduce the viral load, modulate the levels of IgG/IgM, and positively modify the fecal microbiota.

300 adults, 18 to 60 years, RTq-PCR positive for SARS-CoV-2, with mild COVID-19, and SpO2 > 90%, living in Mexico city (2,200m over the sea level) will be randomized, after sign of informed consent to receive a combintation of Lactobacillus plantarum CECT 30292, Lactobacillus plantarum CECT 7484, Lactobacillus plantarum CECT 7485 y P. acidilactici CECT 7483 one a day orally or placebo for 30 days.

Clinical severity, lung abnormalities (x-rays), viral load, IgG/IgM levels, and fecal microbiome will be evaluated at COVID-19 research center before randomization. Participants will be invited to remain at home and clinical evolution, temperature, SpO2 will be recorder and reported remotely during the 30 days intervention.

On days 15 and 30, participants will be invited to return to COVID-19 research center to take samples to evaluate evolution of viral load, IgG/IgM and fecal microbiome.

During the 30-days intervention period outcomes such as clinical progression, need of hospitalization, admission to Intensive Care Unit and death will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Women or men, >18y to 60 years
* RTq-PCR to COVID positive
* Presence of cough, fever, dyspnoea, or headache, onset <= 7 days
* Mild severity of COVID-19
* Peripheral Oxygen Saturation (SpO2) >90%
* Able to read, understand and sign the informed consent
* To have at least one family member to collaborate with the follow-up in the clinical findings at beginning and throughout of the study.

Exclusion Criteria:

* Severe Obesity (BMI>40)
* Uncontrolled Type II diabetes (HbA1C >8.0)
* Uncontrolled systolic hypertension (>160mmdeHg)
* Acute pancreatitis
* Chronic diarrhea or constipation
* Inflammatory bowel disease
* Blood clotting disease
* Immunosuppression derived from Cancer, post-transplantation, auto-immune disease or HIV
* Severe and active seasonal allergies
* Pregnancy or lactation
* Glucose 6P-dehydrogenase deficiency
* Regular use of probiotic or antibiotic within 2 weeks before entering the trial
* Severe or uncontrolled Chronic Respiratory Diseases (Asthma, COPD or Cystic Fibrosis)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Severity progression of COVID-19 | 30 days
  Frequency of randomized subjects who progress from mild to moderate or severe COVID-19, or remission, as evaluated by WHO Clinical Progression Scale
Stay at ICU | 30 days
  Length of stay at Intensive Care Unit (ICU)
Mortality ratio | 30 days
  Mortality ratio for all causes related to COVID-19

SECONDARY OUTCOMES:
Viral load | 30 days
  Description of SARS-Cov-2 viral load evaluated by RT-PCR at screening and on days 15 and 30
Lung abnormalities | 30 days
  Frequency of lung abnormalities clasified by severity and measured by x-ray and artificial intelligence
Levels of immunoglobulins | 30 days
  Levels of Immunoglobulin G and Immunoglobulin M evaluated on day 15 and 30
Gastrointestinal manifestations, where 0 means good health status and 5 worse status | 30 days
  Frequency and severity of gastrointestinal manifestation evaluated by Gastrointestinal Symptom Rating Scale (GSRS)
Fecal microbiome | 30 days
  Changes on fecal microbiome evaluated by 16S analysis on day 1st and 30th
Adverse events | 30 days
  Frequency of adverse events reported on dairy report form after randomization and until day 30
Change on Serum Biomarkers | Days 1st, 15th and 30th after randomization
  Change on high sensitivity C-reactive protein (hsCRP) and D-Dimer
Duration of Individual Symptoms | 30 days
  Days of fever, cough, myalgia, dyspnea and headache

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual patient data (IPD), together with data dictionary defining each field in the set, will be made public upon any formal requests with a defined analysis plan.
Time Frame: From the moment of manuscript publication, without time limit.
Access Criteria: Formal request with a defined analysis plan. Please contact espadaler@ab-biotics.com or medical@ab-biotics.com

REFERENCES:
- [Background] Zuo T, Liu Q, Zhang F, Lui GC, Tso EY, Yeoh YK, Chen Z, Boon SS, Chan FK, Chan PK, Ng SC. Depicting SARS-CoV-2 faecal viral activity in association with gut microbiota composition in patients with COVID-19. Gut. 2021 Feb;70(2):276-284. doi: 10.1136/gutjnl-2020-322294. Epub 2020 Jul 20. PMID 32690600
- [Result] Bottari B, Castellone V, Neviani E. Probiotics and Covid-19. Int J Food Sci Nutr. 2021 May;72(3):293-299. doi: 10.1080/09637486.2020.1807475. Epub 2020 Aug 12. PMID 32787470
- [Result] Klann E, Rich S, Mai V. Gut Microbiota and Coronavirus Disease 2019 (COVID-19): A Superfluous Diagnostic Biomarker or Therapeutic Target? Clin Infect Dis. 2021 Jun 15;72(12):2247-2248. doi: 10.1093/cid/ciaa1191. No abstract available. PMID 32780788
- [Result] d'Ettorre G, Ceccarelli G, Marazzato M, Campagna G, Pinacchio C, Alessandri F, Ruberto F, Rossi G, Celani L, Scagnolari C, Mastropietro C, Trinchieri V, Recchia GE, Mauro V, Antonelli G, Pugliese F, Mastroianni CM. Challenges in the Management of SARS-CoV2 Infection: The Role of Oral Bacteriotherapy as Complementary Therapeutic Strategy to Avoid the Progression of COVID-19. Front Med (Lausanne). 2020 Jul 7;7:389. doi: 10.3389/fmed.2020.00389. eCollection 2020. PMID 32733907
- [Result] De Maio F, Posteraro B, Ponziani FR, Cattani P, Gasbarrini A, Sanguinetti M. Nasopharyngeal Microbiota Profiling of SARS-CoV-2 Infected Patients. Biol Proced Online. 2020 Jul 25;22:18. doi: 10.1186/s12575-020-00131-7. eCollection 2020. PMID 32728349
- [Result] Villena J, Kitazawa H. The Modulation of Mucosal Antiviral Immunity by Immunobiotics: Could They Offer Any Benefit in the SARS-CoV-2 Pandemic? Front Physiol. 2020 Jun 16;11:699. doi: 10.3389/fphys.2020.00699. eCollection 2020. PMID 32670091
- [Result] Marcialis MA, Bardanzellu F, Fanos V. Microbiota and Coronavirus Disease 2019. Which Came First, the Chicken or the Egg? Clin Infect Dis. 2021 Jun 15;72(12):2245-2246. doi: 10.1093/cid/ciaa965. No abstract available. PMID 32645713
- [Result] Aktas B, Aslim B. Gut-lung axis and dysbiosis in COVID-19. Turk J Biol. 2020 Jun 21;44(3):265-272. doi: 10.3906/biy-2005-102. eCollection 2020. PMID 32595361